CLINICAL TRIAL: NCT03200561
Title: A Randomized Open-label Trial to Evaluate the Efficacy of Immunoglobulin Plus Steroid for Prevention of Coronary Artery Abnormalities in Taiwanese Refractory Kawasaki Disease (RAST Study)
Brief Title: A Trial to Evaluate the Efficacy of Immunoglobulin Plus Steroid for Prevention of Coronary Artery Abnormalities in Taiwanese Refractory Kawasaki Disease (RAST Study)
Acronym: RAST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201308036MIND
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Kawasaki Disease; Steroid; Immuoglobulin
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Prednisolone; Immunoglobulins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S group (Active Comparator): IVIG (2g/Kg in 12 hours)+oral prednisolone (2mg/Kg/day for 5 days)
  Interventions: Drug: Prednisolone; Biological: immunoglobulin
- I group (Placebo Comparator): IVIG (2g/Kg in 12 hours)
  Interventions: Biological: immunoglobulin

INTERVENTIONS:
Drug: Prednisolone — Prednisolone 2mg/Kg/day for 5 days
  Arms: S group
Biological: immunoglobulin — immunoglobulin 2g/Kg for 12 hours

SUMMARY:
Background:

Kawasaki disease (KD), most popular acquired heart disease in childhood, is characterized by diffuse vasculitis, especially on the middle-sized muscular arteries. IVIG and aspirin are currently standard treatment. However, 10-15% of KD patients have poor response to such treatment and suffer from higher risk of coronary involvement. Recently, combination of prednisolone and IVIG has been shown effective to lower the chance of refractory to IVIG treatment and subsequent coronary lesions. However, no randomized trial on the steroid efficacy was ever conducted in Taiwan.

Aim:

Prospectively randomized open-label trial to evaluate the add-on effect of prednisolone in the refractory KD children.

Methods:

For the KD patients with fever persisted or relapsed 24 hours after the ending of IVIG infusion, they will be randomized into two group: IVIG group (I) and IVIG + prednisolone group (P). The KD patients in the P group will have in addition to IVIG, oral prednisolone 2mg/kg/day for at least 5 days. The difference in the response rate and percentage of coronary involvement will be compared between I and P groups.

Predicted results:

We plan to enroll 100 refractory KD patients, 50 patients for each group. We predict the risk of coronary involvement can be reduced from 30% to 15%.

ELIGIBILITY:
Inclusion Criteria:

* KD (Kawasaki disease) patients who failed to respond to the initial IVIG as those who had persistent fever that lasted for more than 24 hours (nonresponse to the initial IVIG) or recrudescent fever associated with KD symptoms after an afebrile period (relapse).

Exclusion Criteria:

* KD patients, those diagnosed on or after day 9 of illness (the first illness day was defined as the day of fever onset), those with coronary artery abnormalities before enrolment, those who were afebrile before enrolment, those who had received steroids (oral, intravenous, intramuscular, or subcutaneous) in the 30 days before the study or intravenous immunoglobulin in the previous 180 days, those with concomitant severe medical disorders (eg, immunodeficiency, chromosomal anomalies, congenital heart diseases, metabolic diseases, nephritis, collagen diseases), and those with suspected infectious disease, including sepsis, septic meningitis, peritonitis, bacterial pneumonia, varicella, and influenza.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
maximal coronary z score | one month
  echocardiography

SECONDARY OUTCOMES:
fever more than 38 degree | 3 days
  from end of second course of IVIG

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tai Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan; Mei-Hwan Wu, MD, PhD, Study Director — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Kobayashi T, Kobayashi T, Morikawa A, Ikeda K, Seki M, Shimoyama S, Ishii Y, Suzuki T, Nakajima K, Sakamoto N, Arakawa H. Efficacy of intravenous immunoglobulin combined with prednisolone following resistance to initial intravenous immunoglobulin treatment of acute Kawasaki disease. J Pediatr. 2013 Aug;163(2):521-6. doi: 10.1016/j.jpeds.2013.01.022. Epub 2013 Feb 26. PMID 23485027